CLINICAL TRIAL: NCT03677089
Title: ECHO Autism Replication: Step Wedge Randomized Trial
Brief Title: Extension for Community Healthcare Outcomes Autism Replication Evaluation
Acronym: ECHO Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Toronto (Other); Children's Hospital of Philadelphia (Other); University of Pittsburgh (Other); University of Rochester (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Arkansas (Other); Nationwide Children's Hospital (Other); Vanderbilt University Medical Center (Other); University of California, Irvine (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Karen Kuhlthau, Associate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000415; UA3MC11054 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2018-08-14; First posted 2018-09-19 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism; Telehealth; Primary Care Providers
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Sites were randomized in a stepped-wedge design with 5 clusters (2 sites per cluster) and a staggered start over a 1-year period. Staggering the start allowed for some control for potential temporal trends, as well as allowing the core team to focus on working with each site to ensure smooth startup of the training program at each site.
  All participants received the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECHO Cohort (Experimental): Sites undergo 12 ECHO Autism telehealth clinics. Clusters of two sites each will initiate intervention with 3 months between the start of each cluster.
  Interventions: Behavioral: 12 ECHO Autism telehealth clinics

INTERVENTIONS:
Behavioral: 12 ECHO Autism telehealth clinics — Twice-monthly 2-hour ECHO Autism Clinics will be provided during a 6-month period. Each Clinic will include a didactic presentation, 2 to 3 Primary Care Provider-generated case presentations, expert feedback, and group discussion. Although the ECHO Clinic will include discussion of specific cases, no identifiable personal health information will be shared, individual patients will not be identified, and no direct patient care will be provided.

SUMMARY:
ECHO Autism was intended to assess rigorously the impact of a 12-session telemedicine training program on participating Primary Care Providers (PCP) knowledge, clinical behavior, and self-efficacy in the screening and care of children with Autism Spectrum Disorder (ASD). Each session is referred to as an "ECHO clinic".

DETAILED DESCRIPTION:
The study involved 10 sites (each referred to as an "ECHO Autism Hub"), each running a 12-session training program using a common curriculum and core lecture, with each site expected to recruit 15 PCPs. Sites were randomized in a stepped-wedge design with 5 clusters (2 sites per cluster) and a staggered start over a 1-year period. Staggering the start allowed for some control for potential temporal trends, as well as allowing the core team to focus on working with each site to ensure smooth startup of the training program at each site.

Outcomes are measured at baseline (Month 0), during the intervention (approximately 3 months after the start of the intervention) and after the end of the intervention (approximately 6 months after the start of the intervention). An additional measurement was made 3 months after the end of the intervention to assess whether deterioration occurs after clinic participation ends.

All participants received the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current practice as a primary care provider (PCP)
* Currently providing care for children
* Professional training in: general pediatrics, family medicine, advance practice nursing (i.e. nurse practitioner or physician assistant)
* Active medical license in the state of practice
* Patient population is at least 50% underserved

Exclusion Criteria:

* Trainee status (e.g., medical student, intern, resident, or other pre-professional trainee)
* Subspecialist (e.g., psychiatrists, neurologists, developmental and behavioral pediatricians)
* Practicing within the same practice as another PCP participant (i.e., only one PCP participant from any given practice may be enrolled as a research participant in the study)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Sohl, MD, FAAP, Principal Investigator — University of Missouri Health Care, Thompson Center for Autism; Micah Mazurek, PhD, Principal Investigator — University of Virginia, Curry School of Education

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazurek MO, Parker RA, Chan J, Kuhlthau K, Sohl K; ECHO Autism Collaborative. Effectiveness of the Extension for Community Health Outcomes Model as Applied to Primary Care for Autism: A Partial Stepped-Wedge Randomized Clinical Trial. JAMA Pediatr. 2020 May 1;174(5):e196306. doi: 10.1001/jamapediatrics.2019.6306. Epub 2020 May 4. PMID 32150229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target enrollment was 150. 149 participants, primary care physicians, were screened from 10 ECHO Autism Hub Centers. 1 participant failed screening. 148 participants were enrolled. Screenings/enrollment occurred between September 12, 2016 and January 16, 2018. Two ECHO Autism Hub Centers were randomized to each of the 5 cohorts/clusters.
Pre-assignment Details: The 10 sites were randomly assigned to cohort using SAS. Each site was assigned a random number (from a uniform distribution), and the two lowest numbers were assigned to period 1, etc. through the two highest numbers assigned period 5. No blocking or stratification was used in the randomization.
Groups:
- ECHO Cohort: Cohorts are composed of 12 ECHO Autism telehealth clinics. Clusters of two sites each will initiate intervention with 3 months between the start of each cluster.
Period: Overall Study
Arm/Group | ECHO Cohort
Started | 148
Baseline/Pre-Intervention (5 participants attended but did not complete forms.) | 137
Mid-Intervention | 120
Post-Intervention | 117
Follow-Up | 114
Completed | 114
Not Completed | 34

BASELINE CHARACTERISTICS:
Arm/Group | ECHO Cohort
Number analyzed (Participants) | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 124
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 124
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 21
  Race: Black / African-American | 7
  Race: Other/Multiracial | 4
  Race: White or Caucasian | 100
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114
  Canada | 18

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Pattern of ASD Screening in PCP Charts
Description: Clinical Practice/Behavior for ASD screening will be assessed at four time points by review of a subset of charts from each Primary Care Provider's practice. Four subsets of charts will be reviewed for appropriate ASD screening occurring during well-child visits. Data will be summarized into the percent of children appropriately screened for ASD by each PCP.
Time Frame: Baseline (Month 0), mid-intervention (Month 3), post-intervention (Month 6), and end of follow-up (Month 9)
Population: Participants were not included if they were at the Canadian site because Canadian screening practices are different from the AAP recommendations used in the study. In addition, participants can be included in this outcome measure only if they have children with a well-child visit at 18 or 24 months in the 30 days prior to the chart review.
Measure: Mean (Standard Deviation); unit: percentage of children screened
Groups:
- Baseline: Month 0
- Mid-Intervention: Month 3
- Post-Intervention: Month 6
- End of Follow-Up: Month 9
Arm/Group | Baseline | Mid-Intervention | Post-Intervention | End of Follow-Up
Number analyzed (Participants) | 86 | 86 | 87 | 86
percentage of children screened | 61 (41) | 64 (41) | 66 (40) | 64 (39)

2. Primary Outcome: Longitudinal Pattern of Reported Co-occurring Medical Conditions Correctly Treated in PCP Charts
Description: Clinical Practice/Behavior for treating co-occurring medical conditions will be assessed at four time points by review of a subset of charts from each Primary Care Provider's practice. All visits with an ASD will be reviewed. Data will be summarized into the percent of co-occurring medical conditions appropriately treated by each PCP.
Time Frame: Baseline (Month 0), mid-intervention (Month 3), post-intervention (Month 6), and end of follow-up (Month 9)
Population: Participants can be included in this outcome measure only if they have children with ASD seen in the 60 days prior to the chart review with an identified medical co-morbidity.
Measure: Mean (Standard Deviation); unit: percentage of co-morbid medical problems
Arm/Group | Baseline | Mid-Intervention | Post-Intervention | End of Follow-Up
Number analyzed (Participants) | 69 | 74 | 72 | 72
percentage of co-morbid medical problems | 81 (27) | 76 (30) | 78 (31) | 86 (25)

3. Secondary Outcome: Longitudinal Pattern of Scores on Provider ASD Knowledge Assessment
Description: ASD knowledge will be assessed at four time points using a 33-item unpublished test developed specifically for the current study. The test assesses knowledge in the areas of ASD screening/identification, psychiatric co-morbidities, medical co-morbidities, and management of additional ASD-specific needs.
  This test scores are based on the total number of correct answers, among all 33 questions. Any missing answers are counted as incorrect responses. Scores range from 0-100 with higher scores showing more knowledge of ASD.
Time Frame: Baseline (Month 0), mid-intervention (Month 3), post-intervention (Month 6), and end of follow-up (Month 9)
Population: Participant numbers are based on the number of participants completing the appropriate form at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Baseline | Mid-Intervention | Post-Intervention | End of Follow-Up
Number analyzed (Participants) | 104 | 98 | 103 | 98
score on a scale (0-100) | 49 (22) | 53 (24) | 56 (25) | 57 (26)

4. Secondary Outcome: Longitudinal Pattern of Scores on Provider ASD Self-Efficacy Assessment
Description: Self-Efficacy will be assessed at four time points using a 57-item unpublished questionnaire developed for a previous ECHO Autism pilot study.
  The questionnaire is comprised of five domains: ASD screening and identification, ASD referral and resources, assessment and treatment of medical comorbidities, assessment and treatment of psychiatric comorbidities, and other items. Primary Care Providers report the degree to which they are confident in their ability to provide effective care in each domain. Items are rated on a 6-point Likert-type scale, where 1 = "no confidence" and 6 = "highly confident/expert". Items are summed for a total score and five sub-scale scores. A subscale is marked as missing if more than 20% of responses are missing and the total score is marked as missing if any subscale is marked as missing or if 6 or more of the 57 questions have missing responses. These scores are then normalized to a percentage. Higher scores indicate greater perceived self-efficacy.
Time Frame: Baseline (Month 0), mid-intervention (Month 3), post-intervention (Month 6), and end of follow-up (Month 9)
Population: Participant numbers are based on the number of participants completing the appropriate form at the time points.
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Baseline | Mid-Intervention | Post-Intervention | End of Follow-Up
Number analyzed (Participants) | 104 | 100 | 103 | 98
score on a scale (0-100) | 43 (12) | 61 (11) | 70 (12) | 71 (12)

5. Secondary Outcome: Longitudinal Pattern of the Number of Perceived Barriers to Care
Description: Perceived barriers to caring for children with autism in primary care will be assessed by participant response to an unpublished 9-item checklist and an open response "other" category for a total of 10 possible barriers. A maximum of 10 barriers can be reported and a minimum of 0. More reported barriers indicate more barriers to care.
Time Frame: Baseline (Month 0), mid-intervention (Month 3), post-intervention (Month 6), and end of follow-up (Month 9)
Population: Participant numbers are based on the number of participants completing the appropriate form at the time points.
Measure: Mean (Standard Deviation); unit: reported barriers (count out of 10)
Arm/Group | Baseline | Mid-Intervention | Post-Intervention | End of Follow-Up
Number analyzed (Participants) | 104 | 100 | 104 | 98
reported barriers (count out of 10) | 4.8 (1.6) | 3.7 (1.9) | 2.6 (1.4) | 2.6 (1.5)

6. Secondary Outcome: Participant Satisfaction With ECHO Autism Program
Description: Participant satisfaction will be assessed using an unpublished 12-item survey developed for a previous ECHO Autism pilot study. The survey includes 10 questions assessing overall satisfaction with participation in the ECHO Autism clinic (rated on a 5-point Likert-type scale), and two questions asking for overall comments and suggestions. Participant satisfaction is defined as the percentage of participants who answer 2 = "agree" or 1 = "strongly agree" to question 1 ("Participation in ECHO Autism improved my ability to care for children with autism in my practice").
Time Frame: At end of intervention (Month 6)
Population: Participant numbers are based on the number of participants completing the appropriate form at the time point.
Measure: Number; unit: percentage of of satisfied participants
Arm/Group | ECHO Cohort
Number analyzed (Participants) | 102
percentage of of satisfied participants | 96

7. Secondary Outcome: PCP ECHO Program Attendance
Description: Percentage of the average number of sessions (out of 12) that the participant attended, of those who have completed the program.
Time Frame: At end of intervention (Month 6)
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | ECHO Cohort
Number analyzed (Participants) | 104
percentage of sessions attended | 83 (17)

8. Secondary Outcome: Number of Co-morbidities in Children With ASD
Description: The summary measure is defined as the mean number of co-morbidities reported among the four co-morbidities of interest for a child with ASD. Participants can be included in this outcome measure only if they have children with ASD seen in the 60 days prior to the chart review with an identified medical co-morbidity.
Time Frame: Baseline (Month 0), mid-intervention (Month 3), post-intervention (Month 6), and end of follow-up (Month 9)
Population: Participant numbers are based on the number of participants completing the appropriate form at the time points.
Measure: Mean (Standard Deviation); unit: number of co-morbid conditions per child
Arm/Group | Baseline | Mid-Intervention | Post-Intervention | End of Follow-Up
Number analyzed (Participants) | 91 | 88 | 92 | 95
number of co-morbid conditions per child | 0.67 (0.64) | 0.76 (0.63) | 0.59 (0.55) | 0.68 (0.74)

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | ECHO Cohort
All-Cause Mortality (participants affected / at risk) | 0/132
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT03677089/Prot_000.pdf
  • Statistical Analysis Plan: Original (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03677089/SAP_001.pdf
  • Statistical Analysis Plan: Amendment 1 (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03677089/SAP_002.pdf
  • Statistical Analysis Plan: Amendment 2 (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03677089/SAP_003.pdf